CLINICAL TRIAL: NCT01884480
Title: A Retrospective Analysis of Renal Function, Tac Dose Adjustments and CYP3A5 Pharmacogenetics in Stable Renal Transplant Recipients Converted From Tac BID to Tac OD
Brief Title: Renal Function and Pharmacogenetics in Renal Transplant Recipients Converted From Tac BID to Tac OD
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: FK17
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Real Function Post Conversion From Prograf to Advagraf; Examin Ethnicity and Pharmacogenetics of the Cohort Requiring Dose Adjustment Post-conversion
Keywords: Advagraf, pharmacogenetics, Cyp3A5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 500 Stable renal transplant recipients: cohort of 500 stable RTRS. A subset of this group who required dose adjustment after conversion will be compared to a matched cohort not requiring dose adjustment. Genotyping for Cyp3A5 will be done for both cohorts
- 500 renal transplant recipients: 500 Stable renal transplant recipients converted from prograf to advagraf

SUMMARY:
In Kidney transplant recipients Once daily Tacrolimus has the poteb]ntial advantage of better adnerence, and perhpas improvement in reanl function compred with the twice daily tacrolimus formulation.

Our center has the largest experience in North America with once-daily tacrolimus ( advagraf) in Renal transplant recipients.

Recently we converted ~500 stable patients from the twice daily to once-daily tacrolimus.

We are interested in:

1. change in renal function
2. dose changes based on ethnic diveristy
3. dose changes based on pharmacogenetics

This will helpnus understand better ways to utilize this anti-rejection medication

DETAILED DESCRIPTION:
The Renal transplant program at St. Michael's is one of the largest in Canada. The CNI of choice since 2000 has been tacrolimus based therapy. In 2009 our program decided to switch from bid prograf to once daily advagraf for all de-novo renal transplant recipients (RTR). Our Advagraf experience is currently the largest in North America. Because of concerns regarding generic prograf, we began a conversion of > 600 prevalent transplant patients on bid prograf to OD advagraf in January 2012. At present this is nearly completed.

It has been recognized that dosing of tacrolimus is highly dependent on pharmacogenentic differences related to the CYP3A5 genotype. CYP3A%*3 (nonexpressors) require significantly higher doses of tacrolimus than CYP3A5*1 (expressers) with heterozygotes being somewhere in the middle. Our study will examine the demographics, renal function and tacrolimus dosing and Co levels, both pre and post conversion from tac BID, to tac OD in our cohort of converted patients.

Of More scientific interest, will be to retrospectively determine the CYP3A5 genotypes in recipients who required significant dose adjustments in the tac OD following conversion and compare to a matched cohort of recipients in whom no dose adjustment was needed.

The hypothesis is that recipients who require dose increase when converted from the BID to the OD formulation, will have a different CYP3A5 genotype and will tend towards CYP3A5*3.

This will be the largest cohort to look at this question. Specifically this may lead to better dosing of tac OD, if pre-emptive genotyping prior to transplantation were to be employed.

ELIGIBILITY:
Inclusion Criteria: Renal transplamnt recipients on prograf converted to advagraf

-

Exclusion Criteria:

* none

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 stable renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Difference in Cyp3a5 genotype in recipients requiring dose adjustment in converion from prograf to advagraf | 12 months

SECONDARY OUTCOMES:
change in renal function after conversion from prograf to advagraf | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St.Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Zaltzman AS, Glick LA, Zaltzman JS, Nash M, Huang M, Prasad GV. The role of CYP3A5 polymorphism and dose adjustments following conversion of twice-daily to once-daily tacrolimus in renal transplant recipients. Transplant Res. 2016 Jan 28;5:2. doi: 10.1186/s13737-016-0031-6. eCollection 2016. PMID 26823971